CLINICAL TRIAL: NCT00187057
Title: Pilot Study I for Treatment of Cancer in Children With Ataxia-Telangiectasia
Brief Title: Study for Treatment of Cancer in Children With Ataxia-telangiectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Ataxia-Telangiectasia
Keywords: Ataxia; alphafetoprotein
MeSH Terms: conditions — Ataxia Telangiectasia; Ataxia | interventions — Vinblastine; Vincristine; Prednisone; Daunorubicin; Doxorubicin; Methotrexate; Cyclophosphamide; Asparaginase; Etoposide; Cytarabine; Mercaptopurine; Dexamethasone; Procarbazine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Other): Acute Lymphoblastic Leukemia (ALL) Low Risk
  Interventions: Drug: vinblastine, vincristine, prednisone, daunorubicin; Drug: doxorubicin, methotrexate, cyclophosphamide, L-asparaginase; Drug: etoposide, cytarabine, mercaptopurine; Drug: dexamethasone, procarbazine; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy
- 2 (Other): Acute Lymphoblastic Leukemia (ALL) - High Risk
  Interventions: Drug: vinblastine, vincristine, prednisone, daunorubicin; Drug: doxorubicin, methotrexate, cyclophosphamide, L-asparaginase; Drug: etoposide, cytarabine, mercaptopurine; Drug: dexamethasone, procarbazine; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy
- 3A (Other): B-Cell Non-Hodgkins Lymphoma (Group A)
  Interventions: Drug: vinblastine, vincristine, prednisone, daunorubicin; Drug: doxorubicin, methotrexate, cyclophosphamide, L-asparaginase; Drug: etoposide, cytarabine, mercaptopurine; Drug: dexamethasone, procarbazine; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy
- 3B (Other): B-Cell Non-Hodgkins Lymphoma (Group B)
  Interventions: Drug: vinblastine, vincristine, prednisone, daunorubicin; Drug: doxorubicin, methotrexate, cyclophosphamide, L-asparaginase; Drug: etoposide, cytarabine, mercaptopurine; Drug: dexamethasone, procarbazine; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy
- 4 (Other): Hodgkins Disease
  Interventions: Drug: vinblastine, vincristine, prednisone, daunorubicin; Drug: doxorubicin, methotrexate, cyclophosphamide, L-asparaginase; Drug: etoposide, cytarabine, mercaptopurine; Drug: dexamethasone, procarbazine; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy

INTERVENTIONS:
Drug: vinblastine, vincristine, prednisone, daunorubicin — See Detailed Description section for details of treatment interventions.
Drug: doxorubicin, methotrexate, cyclophosphamide, L-asparaginase — See Detailed Description section for details of treatment interventions.
Drug: etoposide, cytarabine, mercaptopurine — See Detailed Description section for details of treatment interventions.
Drug: dexamethasone, procarbazine — See Detailed Description section for details of treatment interventions.
Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy — See Detailed Description section for details of treatment interventions.

SUMMARY:
This is a pilot/feasibility study designed to investigate the feasibility of treating children with Ataxia-Telangiectasia (A-T) and cancer with regimens nearly as intense as non-A-T patients with cancer would receive.

DETAILED DESCRIPTION:
Approximately 10-30% of A-T patients will develop a malignancy during their lifetime. The vast majority of these cancers are of lymphoid origin. There is no consensus regarding the optimal strategy for treating children with A-T who develop hematopoietic malignancies. Historically, many of these children have been treated with therapy that is much less intensive than the conventional approach for non-A-T patients with similar malignancies during the corresponding treatment era. Although these less intensive approaches may have stemmed from perceptions that these children would not tolerate intensive therapy, there is in fact no data to suggest that these children cannot tolerate intensive therapy. However, it is clear that children with A-T require a modification in certain components of intensive therapy.

To provide children with A-T and either ALL or malignant lymphoma the best chance for a cure, we propose to use modern therapeutic strategies with minimal modifications which address the unique toxicity profile encountered in treating children with A-T.

Secondary objectives include:

* To clinically and biologically characterize the malignancies occurring in children with A-T (usually malignant lymphoma or ALL). This will include in vitro drug sensitivity screening.
* To study chemotherapy-induced DNA damage in children with A-T.

Detailed Description of Treatment Plan:

* Acute Lymphoblastic Leukemia (ALL) Low Risk:

Induction:

Prednisone 40 mg/m2/day PO days 1-28

Vinblastine 6 mg/m2/dose IV day 8

Vincristine 1.5 mg/m2/dose days 1, 15

Daunomycin 20 mg/m2/week IV days 1,15

Asparaginase 10,000 U/m2/dose IM days 2, 4, 6, 8, 10, 12

VP-16 225 mg/m2/dose Days 22, 25, 29

Ara-C 300 mg/m2/dose Days 22, 25, 29

All patients will receive CNS therapy with triple intrathecal therapy on days 1, 22 and 43 of induction treatment, dose age adjusted.

Consolidation:

Methotrexate 2 mg/m2 IV day 43 and 50 and mercaptopurine 75 mg/m2 days 43-56.

Continuation therapy (120 weeks):

Week:

1. 6-MP + MTX
2. 6-MP + MTX
3. 6-MP + MTX
4. Dex + VCR
5. 6-MP + MTX
6. 6-MP + MTX
7. 6-MP + HDMTX
8. Dex + VCR
9. 6-MP + MTX
10. 6-MP + MTX
11. 6-MP + MTX
12. Dex + VCR
13. 6-MP + MTX
14. 6-MP + MTX
15. 6-MP + HDMTX

This sequence will be repeated through week 52 after which 6-MP + MTX will be given weekly to complete 120 weeks. IT MHA (MTX, hydrocortisone, Ara-C) on weeks 1, 2, 7, and 15 and then every 4-8 weeks depending on CNS status.

Dosages, Schedules and Routes:

6-MP 75 mg/m2 PO; daily x 7

MTX 40 mg/m2 IM or IV; q (every) week;

Dex 6 mg/m2 PO; in 3 divided doses daily x 7

VCR 1.5 mg/m2 IV (max. 2.0 mg)

HDMTX 2 g/m2 IV over 2 hours, every 8 weeks

Reinduction:

Reinduction therapy (weeks 16-21). Reinduction therapy (same as initial induction treatment minus dose 2 and 3 of VP16 +ara-C and minus day 22 intrathecal therapy) will be given after bone marrow examination on week 15 confirms complete remission.

* Acute Lymphoblastic Leukemia (ALL) - High Risk

Induction:

Prednisone 40 mg/m2/day PO) divided in 3 doses days 1-28

Vinblastine 6 mg/m2/dose IV day 8

Vincristine 1.5 mg/m2/dose days 1, 15

Daunomycin 20 mg/m2/week IV days 1, 15

Asparaginase 10,000 U/m2/dose IM days 2, 4, 6, 8, 10, 12, (15, 17, 19)

VP16 225 mg/m2/dose days 22, 25, 29

Ara-C 300 mg/m2/dose days 22,25,29

All patients will receive triple IT therapy on days 1, 22 and 43 of induction with additional IT therapy on days 8 and 15 if CNS leukemia (CNS 2 or CNS 3) is present at diagnosis. If required, for patients with CNS 2 and 3 at diagnosis, IT therapy will continue until 2 consecutive CSF studies are normal (i.e., days 29 and 36).

Consolidation:

HDMTX 2 mg/m2 IV day 43 and 50

6 MP 75 mg/m2 PO days 43-56

Continuation Therapy (120 weeks):

Week:

1. Dex + VCR
2. VP-16 + CTX
3. 6-MP + MTX
4. MTX + Ara-C
5. Dex + VCR
6. VP-16 + CTX
7. 6-MP + HDMTX
8. 6-MP + MTX
9. Dex + VCR
10. VP-16 + CTX
11. 6-MP + MTX
12. MTX + Ara-C
13. Dex + VCR
14. VP-16 + CTX
15. 6-MP + HDMTX

These sequences will be repeated through week 52, after which 6MP/MTX will be given weekly to complete 120 weeks.

IT MHA (MTX, hydrocortisone, Ara-C) on weeks 1, 2, 7, and 15 and then every 4-8 weeks depending on CNS status and risk status.

Dosages, Schedules and Routes:

VP 16 225 mg/m2 IV once a week

Cyclophosphamide 300 mg/m2 IV (with MESNA) once a week in addition to the 6 hour IV hydration

6-MP 75 mg/m2 PO; daily x 7

MTX 40 mg/m2 IM or IV once a week

Ara-C 300 mg/m2 IV push; once a week

Dex 8 mg/m2/day PO; in 3 divided doses daily x 7

VCR 1.5 mg/m2 IV push (max. 2.0 mg)

HDMTX 2 g/m2 IV over 2 hours; every 8 weeks x 7

* B-Cell Non-Hodgkins Lymphoma

Overview - the chemotherapy regimen used varies with grouping based on extent of disease

Group A

Induction (COPAD x 2 cycles):

Cyclophosphamide 500 mg/m2/day (divided every 12 hour) IV (with MESNA) Day 1, 2, 3

Vincristine 2.0 mg/m2 IV Day 1

Vinblastine 6 mg/m2 IV Day 6

Prednisone 60 mg/m2/day (bid) PO Day 1-5

Adriamycin 50 mg/m2 (over 6 hrs) IV Day 1

G-CSF 5 mcg/kg/day until count recovery.

Group B

COP Induction:

Cyclophosphamide 300 mg/m2 IV (divided every 12 hours) IV (with MESNA) Day 1

Vincristine 1.0 mg/m2 IV Day 1

Prednisone 60 mg/m2/day (divided bid) PO days 1-7

CNS Therapy Intrathecal Day 1 - dose age adjusted

COPAD-M3 Induction x 2 cycles:

Vinblastine 6 mg/m2 IV Day 1

HD MTX 3 mg/m2 IV over 3 hours Day 1 with leucovorin rescue

CNS Therapy intrathecal each age adjusted Day 2, 6

Cyclophosphamide 500 mg/m2/day (second course 1 mg/m2/day) IV (with MESNA) Day 2, 3, 4

Adriamycin 50 mg/m2 IV Day 2

Prednisone 60 mg/m2 (divided bid) PO Day 1-5

G-CSF 5 mcg/kg/day until count recovery

CYM Consolidation x 2 cycles:

HD MTX 3 mg/m2 IV over 3 hours Day 1 with leucovorin rescue

Ara-C 100 mg/m2/day CI/IV (x 5 days) Day 2-6

CNS Therapy intrathecal each age adjusted Day 2 and 7

Maintenance:

Prednisone 60 mg/m2/day (divided bid) PO Day 1-5

HDMTX 3 mg/m2 IV over 3 hours Day 1 with leucovorin rescue

CNS Therapy intrathecal each age adjusted Day 2

Cyclophosphamide 500 mg/m2/day IV (with MESNA) Day 2, 3

Adriamycin 50 mg/m2 IV Day 3

Vincristine 2 mg/m2 IV Day 1

G-CSF 5 mcg/kg/day until count recovery

* Limited Stage Non-Hodgkins Lymphoma

Induction:

Vincristine 2 mg/m2 IV days 1, 22 (maximum dose 2 mg)

Vinblastine 6 mg/m2 IV, day 8

Prednisone 40 mg/m2/day in 3 divided doses x 28 days

Adriamycin 30 mg/m2/day IV over one hour days 1 and 22

Cyclophosphamide 750 mg/m2/day IV days 1 and 22

Triple IT chemotherapy for participants with head and neck primary tumors on days 1, 8, 22. Each dose age adjusted.

Consolidation - start day 43:

Adriamycin 30 mg/m2 by IV

Cyclophosphamide 750 mg/m2

Prednisone 40 mg/m2 in 3 divided doses x 5 days

Vincristine 2.0 mg/m2 (max. 2.0 mg) by IV

Triple IT chemotherapy for head and neck primaries on days 43 and 64.

Maintenance:

Maintenance chemotherapy will be administered only to patients with lymphoblastic lymphoma and will consist of 24 weeks of chemotherapy with oral daily 6-MP and weekly oral methotrexate (and TIT every 6 weeks for patients with head and neck primaries) after induction/consolidation.

* Hodgkins Disease

Participants with favorable disease will receive VAMP chemotherapy:

VAMP chemotherapy doses and schedule:

Vinblastine 6 mg/m2, IV day 1, 15 (maximum dosage: 10 mg)

Adriamycin 25 mg/m2, IV day 1, 15

Methotrexate 20 mg/m2, IV day 1, 15

Prednisone 40 mg/m2 PO day 1-14 divided into 3 daily doses

Repeat cycle every 28 days, total number of cycles = 6 (NO RADIATION THERAPY)

Participants with unfavorable disease will receive VAMP and COP:

VAMP chemotherapy doses (cycles 1, 3, 5, 7)

Vinblastine 6 mg/m2 IV day 1, 15

Adriamycin 25 mg/m2 IV day 1,15

Methotrexate 20 mg/m2 IV day 1, 15

Prednisone 40 mg/m2 (divided into 3 daily doses) PO day 1-14

COP chemotherapy doses (cycles 2, 4, 6, 8)

Cyclophosphamide 600 mg/m2 IV (with MESNA) day 1, 8

Vincristine 1.4 mg/m2 IV day 1,8 (max dose 2 mg)

Procarbazine 100 mg/m2 PO day 1-14

(NO RADIATION THERAPY)

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of Ataxia-Telangiectasia (A-T).
* Patient must have a diagnosis of either acute lymphoblastic leukemia (ALL) or lymphoma (non-Hodgkin lymphoma or Hodgkin's disease).
* Patients with other malignancies (solid tumors, rare malignancies, or relapsed hematopoietic malignancies) will be eligible for the biologic studies of this protocol; they will receive best clinical management chemotherapy.
* Patients do not have to be previously untreated. If prior chemotherapy has already started (up through induction), therapy will be continued according to protocol at a clinically appropriate time point.

Exclusion Criteria:

* Patients who do not have a diagnosis of Ataxia Telangiectasia (A-T).

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2002-09; Primary Completion 2006-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of delivering modified intensive chemotherapy to children with A-T who present with cancer. | The completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: John T. Sandlund, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Sandlund JT, Kastan MB, Kennedy W, Behm F, Entrekin E, Pui CH, Kalwinsky DT, Raimondi SC. A subtle t(3;8) results in plausible juxtaposition of MYC and BCL6 in a child with Burkitt lymphoma/leukemia and ataxia-telangiectasia. Cancer Genet Cytogenet. 2006 Jul 1;168(1):69-72. doi: 10.1016/j.cancergencyto.2005.12.013. PMID 16772123
- See also: St. Jude Children's Research Hospital — http://www.stjude.org